CLINICAL TRIAL: NCT05592717
Title: An Observational Study of YUTIQ (Fluocinolone Acetonide Intravitreal Implant 0.18 mg) for the Management of Chronic Non-infectious Uveitis
Brief Title: A Study of YUTIQ® 0.18 mg Intravitreal Implant for the Management of Chronic Non-infectious Uveitis
Status: Recruiting | Type: Observational
Sponsor: Tianjin Medical University (Other)
Responsible Party: Principal Investigator, Xiaomin Zhang, Principal Investigator, MD, PhD, Tianjin Medical University
Other Study IDs: 2022KY-17
Record Dates: First submitted 2022-10-19; First posted 2022-10-25 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Uveitis; YUTIQ
MeSH Terms: conditions — Uveitis | interventions — Fluocinolone Acetonide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Yutiq group: Patients will receive YUTIQ® 0.18 mg as an intravitreal injection in the designated study eye and will be followed for 36 months after treatment.
  Interventions: Drug: Yutiq
- traditional therapy group: Patients were treated with glucocorticoids alone or glucocorticoids combined with immunosuppressants and were followed for up to 36 months.

INTERVENTIONS:
Drug: Yutiq — YUTIQ® 0.18 mg as an intravitreal injection in the designated study eye.
  Groups: Yutiq group

SUMMARY:
This project is designed to evaluate the efficacy of YUTIQ® 0.18 mg intravitreal implant for the management of chronic non-infectious uveitis.

DETAILED DESCRIPTION:
Approval of the study was obtained from the hospital's ethical committee. The study design and methodology followed the tenets of Declaration of Helsinki. All patients were provided with written informed consent and received a thorough explanation of the use of Yutiq, its potential risks and benefits. This is a monocenter, cohort, observational study evaluating patients with chronic non-infectious uveitis divided into two groups: Yutiq therapy group and traditional therapy group.

For Yutiq therapy group, patients will receive YUTIQ® 0.18 mg as an intravitreal injection in the designated study eye. For the traditional therapy group, patients were treated with glucocorticoids alone or glucocorticoids combined with immunosuppressants. Study participants will be followed for up to 3 years to determine efficacy and side effects.

According to best corrected visual acuity (BCVA), anterior chamber and vitreous inflammation, optical coherence tomography (OCT), change in corticosteroid dose during the study period and so on. The investigators evaluate the anti-inflammatory and reducing relapses effects of Yutiq in treatment of chronic non-infectious uveitis.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female in good general health at 18 to 70 years of age.
2. Presence of unilateral or bilateral non-infectious uveitis affecting the posterior segment
3. Patients have active inflammation before Yutiq treatment. Subject meets at least 1 of the following criteria: 1. ≥1+ anterior chamber cell and/or ≥1+ vitreous haze. 2. Fluorescein angiography demonstrates leakages. 3. OCT images showing the macular edema. 4. The times of relapse in one year are equal to or greater than 3.
4. Steroids and immunosuppressive agents were discontinued within 3 months after Yutiq injection.

Exclusion Criteria:

1. Subject with corneal or lens opacity that precludes visualization of the fundus or that likely requires cataract surgery during the duration of the trial.
2. Subject with a history of neurologic symptoms suggestive of central nervous system demyelinating disease.
3. Prior intravitreal treatment with Retisert®, ILUVIEN®, or YUTIQ® (0.18 mg) within 36 months prior to Day 1.
4. Prior intravitreal treatment with OZURDEX® within 12 weeks prior to Day 1. Prior intravitreal treatment with Triesence® or TRIVARIS™ (triamcinolone) within 12 weeks prior to Day 1.
5. Peri-ocular or subtenon steroid treatment within 12 weeks prior to Day 1.
6. Media opacity precluding evaluation of retina and vitreous (eg, vitreous hemorrhage).
7. Hypersensitivity to any of the ingredients contained in YUTIQ®.
8. Any other systemic or ocular condition which, in the judgment of the Investigator, could make the subject inappropriate for study enrollment.
9. Pregnant or nursing females; females of childbearing potential who are unwilling or unable to use an acceptable method of contraception as outlined in the protocol from at least 14 days prior to Day 1 until the final study visit.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Chronic non-infectious uveitis patients were recruited from the uveitis centre of Tianjin Medical University Eye Hospital
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2023-01-05 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Change In LogMAR Best Corrected Visual Acuity (BCVA) From Baseline to Each Visit. | 12 months
  Participant's best corrected visual acuity was measured using an Early Treatment Diabetic Retinopathy Study (ETDRS) logMAR chart. On the logMAR scale, 0 is equivalent to 20/20 visual acuity, the range of normal vision is considered to be from -0.2 - 0.1; higher values indicate visual impairment.
Recurrence rates | 36 months
  The recurrence rates in Yutiq group and traditional therapy group

SECONDARY OUTCOMES:
Change in Anterior Chamber (AC) Cell Grade From Baseline to Each Visit | 12 months
  Slit lamp examinations were conducted at each visit to assess AC cell count. The number of AC cells observed within a 1 mm × 1 mm slit beam was used to determine the grade according to the Standardization of Uveitis Nomenclature (SUN) criteria:
  Grade 0 = < 1 cell Grade 0.5+ = 1 - 5 cells Grade 1+ = 6 - 15 cells Grade 2+ = 16 - 25 cells Grade 3+ = 26 - 50 cells Grade 4+ = > 50 cells.
Prednisone exposure | 36 months
  Cumulative prednisone dose and/or mean prednisone dose

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Eye Hospital, Tianjin, Tianjin Municipality, China